CLINICAL TRIAL: NCT01754259
Title: Effects of Ranolazine on Coronary Flow Reserve in Symptomatic Patients With Diabetes and Suspected or Known Coronary Artery Disease
Brief Title: Effects of Ranolazine on Coronary Flow Reserve in Symptomatic Diabetic Patients and CAD
Acronym: RAND-CFR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Marcelo F. Di Carli, MD, FACC, Chief, Nuclear Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2012P002537
Record Dates: First submitted 2012-12-12; First posted 2012-12-21 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Diabetes, Type I; Diabetes, Type II; Angina; Coronary Artery Disease
Keywords: type 1 diabetes; type 2 diabetes; exertion angina; suspected CAD; known CAD
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Angina Pectoris; Coronary Artery Disease | interventions — Ranolazine

STUDY DESIGN:
Intervention Model Description: Subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor. Each patient will receive both ranolazine and placebo for 4 weeks, but both the investigator and subject are blinded to the order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Experimental): Subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor. Each patient will receive both ranolazine and placebo for 4 weeks, but both the investigator and subject are blinded to the order.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor. Each patient will receive both ranolazine and placebo for 4 weeks, but both the investigator and subject are blinded to the order.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor. Each patient will receive both ranolazine and placebo for 4 weeks, but both the investigator and subject are blinded to the order.
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor. Each patient will receive both ranolazine and placebo for 4 weeks, but both the investigator and subject are blinded to the order.
  Other Names: Placebo pill
  Arms: Placebo

SUMMARY:
Coronary vascular dysfunction is highly prevalent among patients with known or suspected Coronary Artery Disease (CAD)1, increases the severity of inducible myocardial ischemia (beyond the effects of upstream coronary obstruction)2, and identifies patients at high risk for serious adverse events, including cardiac death1, 3-5. Diabetic patients without known CAD with impaired coronary vascular function show a risk of cardiac death comparable to, and possibly higher, than that for non-diabetic patients with known CAD10. In the setting of increased oxygen demand, coronary vasodilator dysfunction can upset the supply-demand relationship and lead to myocardial ischemia, subclinical left ventricular dysfunction (diastolic and systolic), and symptoms.

The significance of microvascular coronary dysfunction is increasingly recognized as invasive and non-invasive (PET) methods of quantifying CFR become available.

Importantly, current treatment strategies for obstructive CAD, such as percutaneous coronary intervention with angioplasty and stenting, are not helpful in microvascular disease. Similarly, mortality-altering treatments for systolic heart failure, such as angiotensin converting enzyme inhibitors, have not been beneficial in treating diastolic dysfunction.

DETAILED DESCRIPTION:
Ranolazine is a novel anti-anginal agent which inhibits the late sodium current in cardiomyocytes, decreasing sodium and calcium overload. In ischemia, excess of intracellular calcium may impair myocyte relaxation and contribute to ventricular diastolic stiffness, which in turn affects myocardial contractility and perfusion. Ranolazine is FDA-approved for treatment of chronic angina. In three randomized, placebo-controlled trials of patients with stable angina, it was shown to increase exercise time free of angina and ST-segment depression, increase exercise capacity and decrease angina when used in combination with established antianginal agents including diltiazem, amlodipine or atenolol, and reduce the frequency of angina on patients on maximum doses of amlodipine.Similarly, in a large population of patients with acute coronary syndromes, ranolazine also decreased exertional angina symptoms and incidence of arrhythmias, with no effect on mortality. Interestingly, in this same study, it significantly improved hemoglobin A1c and recurrent ischemia in patients with diabetes mellitus, and reduced the incidence of increased hemoglobin A1c in patients without known prior hyperglycemia.

Although the anti-ischemic effect of ranolazine is thought to be mediated in part by increased myocardial blood flow,there is currently limited evidence for such an effect on tissue perfusion. A previous study in women without overt CAD did not detect improved myocardial blood flow after treatment with ranolazine. In that study, however, coronary hyperemia was elicited with adenosine (which uncouples blood flow from cardiac work, and reflects predominantly endothelial-independent vasodilation) rather than exercise, which triggers a more complex interplay between metabolic demand, coronary hemodynamics, and vasodilator response. Thus, there is a need for additional investigation of whether the beneficial effects of ranolazine on exertional symptoms are directly related to improved global tissue perfusion. Such evidence would support the use of ranolazine as an anti-ischemic therapy in the challenging population of symptomatic patients with evidence of microvascular dysfunction without obstructive CAD.

ELIGIBILITY:
Inclusion Criteria

1. type 1 or 2 diabetes mellitus
2. anginal symptoms and/or exertional dyspnea;
3. ability to exercise and achieve an exercise tolerance of at least 3 METS but not higher than 9 METS either on a treadmill or bicycle exercise tolerance test;
4. perfusion sum stress score (SSS) ≤ 6, as assessed by initial PET

Exclusion Criteria

1. patients not fulfilling inclusion criteria
2. patients with evidence of unprotected left main coronary artery stenosis >50%
3. patients with evidence of new obstructive CAD not on optimal medical therapy
4. evidence of angiographic disease and/or inducible myocardial ischemia on stress testing planning to undergo revascularization within the following 3 months
5. history of cardiomyopathy (LVEF <40%) or significant valvular heart disease
6. uncontrolled hypertension (SBP >180 mm Hg at screening)
7. gait instability, lower extremity amputations preventing exercise

9. significant liver dysfunction (LFTs >3x upper limits of normal), including cirrhosis 10. prolonged QT (QTc >450 and >470 ms for men and women, respectively) or concomitant use of drugs that prolong QT interval (including methadone and antiarrhythmics such as sotalol, amiodarone, and quinidine) 11. use of drugs that inhibit CYP3A such as ketoconazole, itraconazole, fluconazole, clarithromycin, erythromycin, diltiazem, verapamil, nefazodone, nelfinavir, ritonavir, lopinavir, ritonavir, indinavir, and saquinavir 12. use of drugs that induce CYP3A such rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, and St. John's wort 13. atrial fibrillation / inability to hold breath for ≥ 10 seconds (in patients in whom CTA will be performed) 14. eGFR < 50 ml/min or end stage renal disease on dialysis 15. allergy to intravenous contrast 16. pregnant or lactating women, or women of childbearing potential not using an acceptable form of birth control (negative pregnancy test also required) 17. inability to fit safely in PET/CT scanner

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Di Carli, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah NR, Cheezum MK, Veeranna V, Horgan SJ, Taqueti VR, Murthy VL, Foster C, Hainer J, Daniels KM, Rivero J, Shah AM, Stone PH, Morrow DA, Steigner ML, Dorbala S, Blankstein R, Di Carli MF. Ranolazine in Symptomatic Diabetic Patients Without Obstructive Coronary Artery Disease: Impact on Microvascular and Diastolic Function. J Am Heart Assoc. 2017 May 4;6(5):e005027. doi: 10.1161/JAHA.116.005027. PMID 28473401

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The order of ranolazine and placebo exposure was randomly assigned in a 1:1 ratio by the Investigational Drug Service at BWH. During the 28-day treatment periods, ranolazine and matching placebo were administered as 500 mg by mouth twice daily for 1 week and increased to 1000 mg by mouth twice daily for 3 weeks, as tolerated.
Groups:
- Ranolazine: subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor.
  Ranolazine: Subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor.
- Placebo: Subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor.
  Placebo Pill: Subject will receive labeled bottles containing tablets with ranolazine 500 mg or a matching placebo provided by the sponsor.
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 23 | 24
Completed | 18 | 18
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 16 | 12 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 16 | 18 | 34
  Black | 4 | 6 | 10
  Asian | 2 | 0 | 2
  Indian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-exercise Coronary Vasodilator Reserve
Description: Change (from baseline) in post-exercise coronary vasodilator reserve, as measured by PET imaging at 4 weeks post randomization. Per-patient global coronary flow reserve (CFR) was calculated as the ratio of absolute MBF at stress over rest for the entire left ventricle. Quantitation of MBF was performed by two operators blinded to patient, treatment period and treatment order.
Time Frame: 4 weeks
Measure: Number; unit: % change
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 23 | 24
% change | -4 | 2

2. Secondary Outcome: Change in LV Diastolic Function
Description: Change (from baseline) in LV diastolic function reflected primarily in mitral annular early diastolic relaxation velocity (E') at 4 weeks post randomization. LV end-diastolic and end-systolic volumes (used to calculate LVEF), left atrial volume, septal and lateral peak early diastolic tissue velocity (e'), septal and lateral peak systolic tissue velocity (s'), and mitral inflow velocity (E) were all measured in accordance with ASE guidelines.
Time Frame: 4 weeks
Measure: Number; unit: % change
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 23 | 24
% change | 1 | -2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through the telephone follow-up on Day 74.
Description: The definition of adverse events and serious adverse events are the same as the clinicaltrials.gov definitions.
Arm/Group | Ranolazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/24
Other Adverse Events (participants affected / at risk) | 12/23 | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=23) | Placebo (N=24)
Fall complicated by non-fatal intracerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) — One serious adverse event occurred during the placebo period [fall complicated by non-fatal intracerebral hemorrhage].
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=23) | Placebo (N=24)
Nausea and Dizziness (Nervous system disorders) | 9 (9) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Renal abnormality (Renal and urinary disorders) | 1 (1) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest pain requiring evaluation (Cardiac disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations for our study include a relatively small cohort size of 47 patients, that our mechanistic trial was not designed to assess clinical outcomes and that our experimental design allowed for inclusion of patients with non-obstructive CAD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No